CLINICAL TRIAL: NCT00481156
Title: Functional Neuroimaging Effects of Cognitive Remediation Training
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: Minnesota Medical Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 0404M58647; CogRehab
Record Dates: First submitted 2007-05-30; First posted 2007-06-01 (Estimated); Last update posted 2018-05-04 (Actual); Status verified 2018-05

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Cognitive Remediation

STUDY DESIGN:
Intervention Model Description: Randomized, placebo-controlled, single-blind. An untreated healthy control group was also included to examine simple retest effects.
Who Masked: Participant
Masking Description: Participants were randomized to computer-based cognitive training or active social-skills groups. Healthy controls (n=9) received no treatment.

ARMS (3):
- Patients: Cognitive Remediation (Experimental): Patients in the cognitive REM condition attended up to 25 h of training in small groups over 4-6 weeks based on the approach to cognitive remediation described by Wexler and Bell (2005). Patients performed tasks designed to train attention and memory from the battery available within a computerized software package (CogPack Marker Software). This training protocol has been shown to improve memory and executive functioning in patients with schizophrenia (Sartory et al, 2005) and tasks chosen were designed to produce improved working memory and attention capacity in the treated group. In addition, patients in the REM group trained on the word N-back one to two times a week and on N-back tasks using a variety of other stimuli (such as faces) one to two times a week to support the generalization of working memory improvements.
  Interventions: Behavioral: Cognitive Remediation
- Patients: Cognitive-Behavioral Social Skills Training (Active Comparator): Patients in the CBSST group also attended up to 25 h of treatment but followed a manualized group therapy protocol (Granholm et al, 2005) using cognitive and behavioral therapy methods to increase patients' skills in symptom recognition, communication, problem solving, and relapse prevention. In both conditions, the facilitators interacted with the clients throughout small group (B4 patients) sessions: in the REM group, this mostly involved brief one-on-one discussions regarding task performance; in the CBSST condition, this interaction was in the context of the group milieu.
  Interventions: Behavioral: Cognitive Behavioral Social Skills Training
- Controls: Retest control group (Other): Estimate of normal brain functioning and retest effects
  Interventions: Other: Retest in Health Controls

INTERVENTIONS:
Behavioral: Cognitive Remediation
  Arms: Patients: Cognitive Remediation
Behavioral: Cognitive Behavioral Social Skills Training
  Arms: Patients: Cognitive-Behavioral Social Skills Training
Other: Retest in Health Controls — Pre/Post test performance and neuroimaging only
  Arms: Controls: Retest control group

SUMMARY:
The purpose of this study is to examine behavioral and functional brain changes occuring as a result of cognitive remediation training in patients with schizophrenia. Extension and specificity of related changes will also be examined.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia or schizoaffective disorder
* Stable outpatient

Exclusion Criteria:

* Current drug abuse or dependence
* History of neurological damage, disorder, or disease

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2005-03-01 (Actual); Primary Completion 2007-02-28 (Actual); Study Completion 2007-02-28 (Actual)

PRIMARY OUTCOMES:
Working Memory performance | Post-test
  N-Back Performance
Brain activation | Post-test
  Changes in prefrontal cortical functioning

CONTACTS AND LOCATIONS:
Overall Officials: Angus W MacDonald, Ph.D., Principal Investigator — University of Minnesota; Kelvin O Lim, Ph.D., Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Haut KM, Lim KO, MacDonald A 3rd. Prefrontal cortical changes following cognitive training in patients with chronic schizophrenia: effects of practice, generalization, and specificity. Neuropsychopharmacology. 2010 Aug;35(9):1850-9. doi: 10.1038/npp.2010.52. Epub 2010 Apr 28. PMID 20428109